CLINICAL TRIAL: NCT06986161
Title: Optimizing Mango's Glycemic Impact: Investigating Mango Consumption Timing in Relation to Meal in Prediabetic Individuals
Brief Title: Optimizing Mango's Glycemic Impact: Investigating Mango Consumption Timing in Prediabetic Individuals
Acronym: MG3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: National Mango Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-95
Record Dates: First submitted 2025-05-07; First posted 2025-05-22 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Mangifera indica extract

STUDY DESIGN:
Intervention Model Description: The pilot study will use a single-blinded, randomized, 4-arm, within-subjects crossover design lasting approximately 5 weeks.
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mango Before Meal (Experimental): 1 cup (165 grams) of mango before standardized breakfast
  Interventions: Other: Mango
- Mango With Meal (Experimental): 1 cup (165 grams) of mango with standardized breakfast
  Interventions: Other: Mango
- Mango After Meal (Experimental): 1 cup (165 grams) of mango after standardized breakfast
  Interventions: Other: Mango
- Control (no mango) (Placebo Comparator): Control beverage (230 grams) with standardized breakfast
  Interventions: Other: Control Beverage

INTERVENTIONS:
Other: Mango — Mango beverage
  Arms: Mango After Meal; Mango Before Meal; Mango With Meal
Other: Control Beverage — Italian Ice beverage
  Arms: Control (no mango)

SUMMARY:
The purpose of this study is to investigate the effect of mango intake on metabolic and inflammatory responses relative to meals in individuals at risk of developing diabetes, as well as to understand how the beneficial compounds found in mangoes are absorbed and processed in the body.

DETAILED DESCRIPTION:
The primary goal of the proposed project is to advance current knowledge about the antidiabetic and anti-inflammatory benefits of consuming mangoes, especially in individuals with prediabetes, and to determine the best timing of mango intake relative to meals.

Participation in this study will last approximately five weeks and will include six visits: one screening visit lasting about one hour and four study-day visits, each lasting approximately eight hours. During these study visits, blood and urine samples will be collected to help researchers better understand the effects of mango intake relative to meal consumption.

Screening Visit:

Participant eligibility for the study is based on the inclusion and exclusion criteria. To assess this, the participant will need to arrive at the Clinical Nutrition Research Center (CNRC) fasting for 10-12 hours, meaning no food or drink other than plain water during this period.

During the screening visit, the following assessments will be conducted:

* The participant will complete a screening questionnaire about their health, dietary habits, and physical activity history.
* The participant's height, weight, waist circumference, and body composition will be measured. Their Body Mass Index (BMI) will be calculated based on their height and weight. BMI is an estimate of body fat that applies to both adult men and women.
* The participant's forehead temperature, blood pressure, and heart rate will be measured. They will be seated in a comfortable chair with their feet flat on the ground and uncrossed. They will be asked to relax for five minutes before their blood pressure and heart rate are recorded.
* A finger prick test will be performed to check their blood sugar levels.
* A licensed healthcare practitioner (LHCP) and/or a certified phlebotomist will assess their arm veins using a vein access scale test. A butterfly needle will then be used to draw 3 milliliters (mL) of blood from their arm to measure their plasma blood glucose levels.
* If the participant is a woman under the age of 60 year, they will be required to take a pregnancy test.

Based on the results of the questionnaire, blood glucose levels, physical measurements, and overall health evaluation, the participant may meet the eligibility criteria and be invited to participate in the study. If eligible, they will also be instructed to complete a 24-hour food recall, documenting their food intake over the past day.

PRE-STUDY VISIT: (which may take place on the same day as the screening visit or on a different day)

If the participant qualifies based on their screening results, the Pre-Study visit can take place immediately after their screening or on a later date. This visit lasts approximately 30-45 minutes, during which they will meet with one of our investigators who will provide detailed instructions on the study procedures and how to prepare for each study day. They will also receive training on study procedures, including dietary restrictions, medications and supplements to avoid, food and gastrointestinal assessment (GI-tract diary recording), and overnight fasting requirements. Their study dates will be scheduled, and they will receive a study booklet containing their study calendar and all the instructions covered during the Pre-Study visit.

Procedures for Each Study Day Visit (Visits 1, 2, 3, and 4)

Participants will visit the Clinical Nutrition Research Center (CNRC) on four separate occasions, with a seven-day washout period between each visit. They will consume either the equivalent of one cup of fresh mango (165 grams, ~100 kilocalories) or a calorie-matched control beverage (230 grams, ~100 kilocalories) before, with, or after a meal, as outlined in the study schema.

Confirmation that the participant is prepared for a study day visit: We will collect their three-day food record and verify that they have fasted overnight, consumed a standardized dinner meal, avoided the specified food items, had sufficient sleep, and maintained dietary and exercise patterns consistent with the study procedures. Once everything is confirmed, they will proceed to an exam room, where we will measure their weight, body composition, vital signs (blood pressure, heart rate, and forehead temperature), and check their fasting blood glucose with a finger prick test.

Urine collection: The participant will collect a urine sample using a urine collection cup at the start of the visit (0 hours). Additional samples will be collected at 1 hour, 2 hours, 3 hours, 5 hours, and 7 hours, for a total of six collections throughout the visit.

Blood collection: The Licensed Health Care Provider (LHCP) will collect their blood samples. They can choose between an intravenous catheter or multiple butterfly sticks. A total of seven blood draws will be taken at 0 hours, 0.5 hours, 1 hour, 2 hours, 3 hours, 5 hours, and 7 hours.

Study Beverages and Standardized Breakfast: Once the fasting blood and urine samples are collected, they will receive a pre-meal study beverage. After the 1-hour blood draw, they will be provided with a standardized breakfast meal and a study beverage. Following the 2-hour blood draw, they will receive a post-meal study beverage.

ASA24 Food Recall: The Online Dietary Questionnaire (ASA24) is a web-based questionnaire. We will ask the participant to report everything they ate and drank over the previous day. This questionnaire may take up to 45 minutes to complete each time.

At the End of the Study Day: The participant will be evaluated for safety and any discomfort or symptoms before leaving. They will receive a take-home snack, and compensation will be issued after all study procedures are completed. Additionally, they will be given instructions on how to prepare for their next visit.

How much blood will be collected during the study visit?: During each of the four study visits, blood will be collected a total of seven times per visit, with a total of 280 milliliters of blood collected throughout the study across all visits.

ELIGIBILITY:
Inclusion Criteria:

* Be between 20-60 years old.
* Have a BMI of 25-35 kilograms per square meter.
* Have fasting blood glucose between 100-125 milligrams per deciliter or Glycated hemoglobin (HbA1c) between 5.7-6.4%.
* Be non-smokers for at least 12 months.
* Be generally healthy, with no major organ-related diseases.
* Not take medications or supplements that could interfere with the study.
* Be able to follow study procedures, including dietary restrictions and scheduled visits.

Exclusion Criteria:

* Smoke, vape, or use marijuana.
* Have allergies or intolerance to mangoes or study foods.
* Have blood pressure above 160/100 millimeters of Mercury.
* Have fasting blood glucose above 125 milligrams per deciliter.
* Have a history of major heart disease, stroke, or cancer in the past five years.
* Be pregnant, planning to become pregnant, or breastfeeding.
* Take anti-inflammatory drugs or certain dietary supplements.
* Have had major surgery or trauma in the past two months.
* Follow extreme diets (e.g., vegan, Atkins).
* Have used antibiotics in the last six weeks.
* Have a history of eating disorders or substance abuse in the past two years.
* Drink more than three cups of coffee or tea per day.
* Have donated blood in the last three months.
* Be professional athletes or do excessive exercise.
* Have had weight changes of more than 11 pounds in the past two months.
* Work overnight shifts.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in postprandial glucose | 7 hours
  Change in postprandial glucose as measured by absolute values and calculated insulin sensitivity using homeostasis model assessment of fasting insulin sensitivity (HOMA-%S) and B-cell function (HOMA-%).
Change in postprandial glucose through peripheral insulin sensitivity | 7 hours
  Change in postprandial glucose as measured by assessment of peripheral insulin sensitivity using Matsuda index.
Change in postprandial insulin | 7 hours
  Change in postprandial insulin as measured by absolute values and calculated insulin sensitivity using homeostasis model assessment of fasting insulin sensitivity (HOMA-%S) and B-cell function (HOMA-%).
Change in postprandial insulin through peripheral insulin sensitivity | 7 hours
  Change in postprandial insulin as measured by assessment of peripheral insulin sensitivity using Matsuda index.
Evaluate Interleukin-6 (IL-6) as an index of systemic inflammatory response | 7 hours
  Assessments to address this aim will include analysis of systemic markers of inflammation (IL-6) in plasma using ELISA method
Evaluate Tumor Necrosis Factor-alpha (TNF-α) as an index of systemic inflammatory response | 7 hours
  Assessments to address this aim will include analysis of systemic markers of inflammation (TNF-α) in plasma using ELISA method

SECONDARY OUTCOMES:
Characterize metabolite profiles | 7 hours
  Polyphenolic metabolites (phenolic acids and derivatives components) will be identified and quantified in urine and plasma. Metabolites in samples will be identified and quantified using an Agilent 6550 iFunnel ultra-high performance liquid chromatography-quadrupole time-of-flight mass spectrometry (UHPLC/Q-TOF-MS) and 6460 ultra-high performance liquid chromatography- triple quadrupole mass spectrometry (UHPLC-QQQ-MS), respectively

CONTACTS AND LOCATIONS:
Overall Officials: Indika Edirisinghe, PhD., Principal Investigator — Illinois Institute of Technology; Britt Burton-Freeman, PhD., Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No